CLINICAL TRIAL: NCT07035522
Title: Evaluation of the Effects of Ozone Therapy on Endometriosis
Brief Title: Ozone Therapy for Women With Endometriosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Collaborators: Philozon Geradores de Ozonio LTDA (Industry)
Responsible Party: Principal Investigator, Henrique Cunha Carvalho, Evaluation of the effects of ozone therapy on endometriosis, Universidade Federal do Paraná
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7.499.295; 86719325.4.0000.0177 (Other: CEP UTFPR)
Record Dates: First submitted 2025-06-02; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis; Ozone Therapy; Thermography
Keywords: ozone; ozone therapy; ultrasound; thermography
MeSH Terms: conditions — Endometriosis | interventions — Thermography; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ozone therapy on endometriosis (Experimental): The participants will undergo anamnesis, including clinical and epidemiological aspects for this research, including the capture of thermographic images. The participants will have previously undergone the transvaginal ultrasound examination; These participants will undergo 10 sessions, within the pre-established protocol with ozone. The selected participants will be allocated into two groups: Group A (ozone therapy) and Group B (control group - conventional treatment). Each group will consist of 20 participants. - Group A (Ozone Therapy): The participants in this group will undergo ozone therapy sessions, according to the established protocol, and will receive treatment in the pelvic cavity with an initial injection of ozonated water, followed by an injection of ozone gas. The application of ozone will be done according to standardized and referenced techniques. - Group B (Clinical treatment): The participants in this group will be monitored to compare the results.
  Interventions: Other: Ozone therapy

INTERVENTIONS:
Other: Ozone therapy — The study also aims to analyze the efficacy of ozone therapy in participants affected by endometriosis, enriching the knowledge base in the field of women's health/gynecology. The expected results will contribute to improving current therapeutic approaches, informing clinical decisions and encouraging future research. Understanding the technique and its clinical applicability will help health professionals to offer personalized and effective treatments. In addition, the insights obtained can direct new investigations, such as the optimization of protocols or the exploration of innovative therapeutic combinations for even more satisfactory results. Based on the literature review and the biochemical properties of both techniques (ozone therapy and clinical approach), it may be possible that one of the approaches demonstrates a statistically superior advantage over the other. In addition, the research aims to investigate whether the quality of life of these participants will improve and i
  Other Names: thermography; ultrasound

SUMMARY:
To evaluate the action of ozone therapy as an adjuvant treatment in patients with endometriosis. Secondary Objective: To evaluate the efficacy of ozone therapy for pelvic analgesia in women with endometriosis; To compare the imaging diagnostic techniques of transvaginal ultrasound with infrared thermography in the pre-treatment (before), fourth, seventh and post-treatment (10th session) periods; To evaluate the application of the consolidated questionnaire (EHP-30) in the changes in the quality of life of the participants immediately after the intervention.

DETAILED DESCRIPTION:
Endometriosis is a chronic gynecological condition characterized by the abnormal presence of endometrial glands and stroma outside the uterus, accompanied by chronic inflammation. It is found mainly in girls and women of reproductive age, and according to data from the World Health Organization, it occurs in approximately 10% of women of reproductive age (190 million) worldwide. Effective management of endometriosis requires rapid diagnosis to allow early multidisciplinary intervention that aligns with the patient's needs and priorities. The etiopathogenesis is not yet well established, but evidence indicates that the combination of genetic, hormonal and immunological factors may contribute to the formation and development of ectopic foci of endometriosis. The clinical picture is quite variable. It may be asymptomatic, refer only to infertility or have symptoms such as severe dysmenorrhea, deep dyspareunia, chronic pelvic pain, ovulatory pain, urinary or perimenstrual evacuation symptoms and chronic fatigue. Uncertainty and delays in diagnosis contribute to disturbances in the emotional system, impacting on quality of life. The objective of this research project is to evaluate the effectiveness of ozone therapy and the assessment by means of diagnostic imaging examinations using transvaginal ultrasound and infrared thermography, before, during and after the intervention, aiming at a comparative investigation of possible evidence of the evolution of patients diagnosed with endometriosis who did not respond to conventional treatments, as well as to apply a consolidated questionnaire that assesses changes in the quality of life of the participants after the intervention. This study is part of an experimental research project and will be carried out in a private clinic, Clínica Fernanda Ferraz - Fisioterapia Integrativa LTDA. The clinic is located at Travessa João Turin, 37, room 603 - Água Verde, Curitiba-PR. The target population of this study will be composed of women between the ages of 25 and 45, with a diagnosis based on a report of endometriosis (all stages will be treated). A convenience sample will be used, recruited through advertisements on social networks. A total of 40 participants will be selected for the study, divided equally into two groups: Group A (ozone therapy) and Group B (control group - conventional clinical treatment). This study will contribute to a deeper understanding of the effects of ozone therapy on endometriosis. It is expected that a statistically significant analysis will be observed that will highlight important differences in imaging in transvaginal ultrasound and thermographic examinations, as well as in symptoms and quality of life. Based on the literature review and the biochemical properties of both techniques (ozone therapy and clinical approach), it is likely that one of the approaches will demonstrate a statistically superior advantage over the other. In addition, the research aims to investigate whether the quality of life of the participants will improve, and in some cases, with potential positive results on infertility.

ELIGIBILITY:
Inclusion Criteria:

* Women with a clinical diagnosis of endometriosis (ultrasonography / transvaginal exam)
* 25-45 years old

Exclusion Criteria:

* Pregnancy
* G6PD positive
* Addicted
* HIV and hepatitis positive
* Cancer
* Anticoagulant sensitive
* Endometrial surgery history

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-18 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
EHP-30 - Endometriosis Health Profile Questionnaire | EHP-30 will be applied at pre (baseline), through study completion, an average of 2 months.
  The EHP-30 (Endometriosis Health Profile-30) is a disease-specific, patient-reported outcome measure designed to assess the health-related quality of life (HRQoL) in individuals with endometriosis on various aspects, including physical, emotional, and social well-being.

SECONDARY OUTCOMES:
Thermographic images | Infra-red images will be captured at pre (baseline), through study completion, an average of 2 months.
  Thermography, a non-invasive imaging technique that detects infrared radiation to map skin surface temperature, will be applied as a tool to assess the physiological response to ozone therapy in endometriosis. Ozone therapy, known for its anti-inflammatory and analgesic properties, may influence local blood flow and immune activity. Thermographic imaging allows visualization of these changes by capturing temperature variations in the abdominal or pelvic regions before (baseline), during (4 and 7th session) and after treatment (10th session). In endometriosis, affected areas often exhibit thermal asymmetry or increased heat due to inflammation. Post-ozone therapy, thermography can reveal reductions in localized hyperthermia, suggesting decreased inflammation and improved circulation. This method provides a visual, quantifiable means to monitor treatment response over time, offering a complementary assessment tool alongside symptom tracking.

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Cunha Carvalho, PhD. Dr., Study Chair — UTFPR
Locations (1):
- Clínica Fernanda Ferraz - Fisioterapia Integrativa LTDA, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
Ethical or Consent Restrictions: Participants may not have given explicit consent for their data to be shared beyond the original study.
  Legal or Institutional Policies: Data sharing may be restricted by Brazillian laws.

REFERENCES:
- [Background] Pires MV, de Lima CJ, Carvalho HC, Moreira LH, Fernandes AB. Effectiveness of intravesical ozone in interstitial cystitis by the O'Leary-Sant symptom index. Int Urogynecol J. 2023 Jul;34(7):1437-1446. doi: 10.1007/s00192-022-05383-3. Epub 2022 Oct 15. PMID 36242631
- [Background] Wei A, Feng H, Jia XM, Tang H, Liao YY, Li BR. Ozone therapy ameliorates inflammation and endometrial injury in rats with pelvic inflammatory disease. Biomed Pharmacother. 2018 Nov;107:1418-1425. doi: 10.1016/j.biopha.2018.07.137. Epub 2018 Sep 1. PMID 30257358
- [Background] Merhi Z, Garg B, Moseley-LaRue R, Moseley AR, Smith AH, Zhang J. Ozone therapy: a potential therapeutic adjunct for improving female reproductive health. Med Gas Res. 2019 Apr-Jun;9(2):101-105. doi: 10.4103/2045-9912.260652. PMID 31249259
- [Background] Gupta S, Goldberg JM, Aziz N, Goldberg E, Krajcir N, Agarwal A. Pathogenic mechanisms in endometriosis-associated infertility. Fertil Steril. 2008 Aug;90(2):247-57. doi: 10.1016/j.fertnstert.2008.02.093. PMID 18672121
- [Background] Nisolle M, Donnez J. Peritoneal endometriosis, ovarian endometriosis, and adenomyotic nodules of the rectovaginal septum are three different entities. Fertil Steril. 1997 Oct;68(4):585-96. doi: 10.1016/s0015-0282(97)00191-x. PMID 9341595
- [Background] Wright CI, Kroner CI, Draijer R. Non-invasive methods and stimuli for evaluating the skin's microcirculation. J Pharmacol Toxicol Methods. 2006 Jul-Aug;54(1):1-25. doi: 10.1016/j.vascn.2005.09.004. Epub 2005 Oct 25. PMID 16256378
- [Background] Horne AW, Saunders PTK. SnapShot: Endometriosis. Cell. 2019 Dec 12;179(7):1677-1677.e1. doi: 10.1016/j.cell.2019.11.033. Epub 2019 Dec 12. PMID 31951524
- [Background] Ahn SH, Singh V, Tayade C. Biomarkers in endometriosis: challenges and opportunities. Fertil Steril. 2017 Mar;107(3):523-532. doi: 10.1016/j.fertnstert.2017.01.009. Epub 2017 Feb 8. PMID 28189296
- [Background] Smolarz B, Szyllo K, Romanowicz H. Endometriosis: Epidemiology, Classification, Pathogenesis, Treatment and Genetics (Review of Literature). Int J Mol Sci. 2021 Sep 29;22(19):10554. doi: 10.3390/ijms221910554. PMID 34638893
- [Background] Saunders PTK, Horne AW. Endometriosis: Etiology, pathobiology, and therapeutic prospects. Cell. 2021 May 27;184(11):2807-2824. doi: 10.1016/j.cell.2021.04.041. PMID 34048704